CLINICAL TRIAL: NCT06766682
Title: The Effect of Skill Development Program for Emotion Regulation on Emotion Regulation, Experiential Avoidance and Compassion Fatigue of Oncology Nurses
Brief Title: Emotion Regulation Skill Program: Impact on Emotion Regulation, Experiential Avoidance & Compassion Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aycan Kayalar, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AYCAN KAYALAR
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Compassion Fatigue; Experiential Avoidance; Emotion Regulation Abilities; Emotion Regulation
Keywords: oncology nursing; difficulty in emotion regulation; emotion regulation skill; experiential avoidance; compassion fatigue
MeSH Terms: conditions — Compassion Fatigue; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Skill Development Program for Emotion Regulation (Experimental): The Skill Development Program for Emotion Regulation to be carried out with the intervention group consists of 6 sessions. The sessions are planned to be held in 3 groups of 11 people. The duration of a session is planned to be 90 minutes. Sessions will be completed in three weeks, twice a week. Sessions will be face-to-face. The session of the same group will be held on the same day and time every week.
  Interventions: Behavioral: The Skill Development Program for Emotion Regulation
- Control Group (No Intervention): After the follow-up tests were completed for the nurses in the control group, the 6-session skill program applied to the intervention group was planned to be applied in the same way within their wishes.

INTERVENTIONS:
Behavioral: The Skill Development Program for Emotion Regulation — The Skill Development Program for Emotion Regulation to be carried out with the intervention group was planned as 6 sessions. The aim of this study was to investigate The Skill Development Program for Emotion Regulation Program on oncology nurses' emotion regulation difficulties, emotion regulation skills, experiential avoidance, and compassion fatigue.
  Arms: The Skill Development Program for Emotion Regulation

SUMMARY:
In this study, the effects of the skills development program for regulating emotions applied to oncology nurses on oncology nurses' emotion regulation, experiential avoidance, and comorbidity fatigue will be examined. The research will be conducted as a randomized controlled experimental study with pretest-posttest and follow-up design.

DETAILED DESCRIPTION:
Cancer has profound emotional, psychological, and behavioral impacts on patients and caregivers. Oncology nurses, while providing care, often experience feelings of helplessness, sadness, anxiety, and anger. Shift work-induced insomnia and irregular living patterns can impair emotional regulation, negatively affecting nurses' ability to provide holistic care, make effective decisions, and maintain professional interactions. Emotional recognition and management skills are critical for nurses engaged in long-term care processes. Emotional regulation involves identifying, understanding, and managing emotional responses, encompassing awareness, appropriate management, and expression. Ineffective emotional regulation may lead to difficulties in coping with emotional challenges and increase the risk of developing disorders such as depression and anxiety.

The literature highlights that emotional regulation strategies, which involve specific skills to modify emotional experiences, play a significant role in the development of various psychopathological disorders and affect mental health. Maladaptive strategies such as experiential avoidance-defined as avoiding situations or thoughts to escape distressing emotions-have been linked to increased risks of anxiety, depression, and burnout. Effective emotional regulation strategies are crucial for maintaining mental health and influencing behaviors. Increased experiential avoidance among healthcare workers has been associated with higher levels of burnout.

Empathy is a cornerstone of psychosocial care for patients and their families in oncology clinics. However, failure to regulate emotions during empathetic interactions can result in compassion fatigue, characterized by physical and emotional exhaustion, anger, disengagement, reduced job performance, and patient dissatisfaction. Effective emotional regulation supports the delivery of empathetic care and protects the psychosocial well-being of nurses. Emotional regulation enhances individuals' emotional awareness and enables more conscious and controlled management of emotions. This study aims to investigate the impact of an emotional regulation skills development program on oncology nurses' emotional regulation difficulties, experiential avoidance, and compassion fatigue in challenging work environments.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Working in the specified units for at least six months
* Not having a disease or disability would make it difficult for them to understand the program and data collection tools and to apply the skills.

Exclusion Criteria:

* Having received or currently receiving individual or group psychotherapy/counseling program within the last six months
* Requesting to withdraw from the study at any stage of the research
* Regularly missing two consecutive group sessions
* Failure to attend three or more sessions in total

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-08-02 (Estimated)

PRIMARY OUTCOMES:
Change in Difficulty in Emotion Regulation Scale-Short Form | [Time Frame: Baseline, 3th week, 3st month follow-up) (Pretest-posttest follow-up experimental design)
  Difficulty in Emotion Regulation Scale-Short Form consists of 16 items and 5 sub-dimensions in 5-point Likert type (1=almost never, 5=almost always). It has five sub-dimensions: Clarity, Goals, Impulse, Strategies, and Non-Acceptance. A minimum score of 16 points and a maximum score of 80 points can be obtained from the scale and high scores obtained from the sub-dimensions and total score of the scale indicate that emotion regulation difficulties are high.

SECONDARY OUTCOMES:
Change in the Emotion Regulation Skills Scale | [Time Frame: Baseline, 3th week, 3st month follow-up) (Pretest-posttest follow-up experimental design)
  The Emotion Regulation Skills Scale is a five-point Likert-type (1=almost never, 5=almost always) self-report instrument consisting of 27 items and nine subscales. The sub-dimensions are Awareness/attention, Body sensations, Clarity, Understanding, Acceptance, Tolerance, Preparation for confrontation, Self-support, and Modification. The minimum score that can be obtained from the scale is 27 and the maximum score is 135. The scale can be evaluated on the total score and the average of the sub-dimension scores

OTHER OUTCOMES:
Change in the Multidimensional Experiential Avoidance Scale-30 | [Time Frame: Baseline, 3th week, 3st month follow-up) (Pretest-posttest follow-up experimental design)
  This scale is a 7-point Likert-type (1: Strongly Disagree; 7: Strongly Agree) self-report instrument consisting of 30 items. The minimum score is 30 points and the maximum score is 210 points. This scale has 6 subscales. These subscales consist of behavioral avoidance, aversion to distress, procrastination, distraction/suppression, suppression/denial and endurance of distress. The increase in the scores obtained from the scale means an increase in the level of the related dimension. Only item 15 of the scale items is reverse scored. However, it is possible to get a total score; however, for this purpose, it is necessary to reverse score the distress tolerance dimension.
Change in the Compassion Fatigue Short Scale | [Time Frame: Baseline, 3th week, 3st month follow-up) (Pretest-posttest follow-up experimental design)
  This scale is a 10-point Likert-type scale ranging from rarely/never (1) to very often (10) and consists of 13 items. The lowest score is 13 and the highest score is 130. As the scores obtained from the scale increase, the level of co-sensory fatigue experienced by individuals also increases. The scale consists of two sub-dimensions: 'secondary trauma' and 'occupational burnout'
Participant Information Form | Time Frame: baseline
  The participant information form included questions about the descriptive characteristics of the nurses. In this context, it includes eight questions such as age, gender, education level, marital status, working time as a nurse, working time as an oncology nurse, number of patients cared for daily, working time per week, place of work, psychiatric diagnosis or treatment, individual or group psychotherapy or psychological counseling program in the past

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU HİÇDURMAZ, Professor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett MD, Hays KN, Cantu C. Compassion fatigue, emotional labor, and emotional display among hospice nurses. Death Stud. 2022;46(2):290-296. doi: 10.1080/07481187.2019.1699201. Epub 2019 Dec 9. PMID 31814533
- [Background] Figley, C. R. (2013). Compassion fatigue: Coping with secondary traumatic stress disorder in those who treat the traumatized. Routledge.
- [Background] Guner P, Hicdurmaz D, Kocaman Yildirim N, Inci F. Psychosocial care from the perspective of nurses working in oncology: A qualitative study. Eur J Oncol Nurs. 2018 Jun;34:68-75. doi: 10.1016/j.ejon.2018.03.005. Epub 2018 Mar 16. PMID 29784141
- [Background] Lincoln, T. M., Schulze, L., & Renneberg, B. (2022). The role of emotion regulation in the characterization, development and treatment of psychopathology. Nature Reviews Psychology, 1(5), 272-286
- [Background] Yiğit, İ. ve Guzey-Yiğit, M. (2019). Psychometric properties of Turkish version of difficulties in emotion regulation scale-brief form (DERS-16). Current Psychology, 38, 1503-1511. https://doi.org/10.1007/s12144-017-9712-7
- [Background] Zheng RS, Guo QH, Dong FQ, Owens RG. Chinese oncology nurses' experience on caring for dying patients who are on their final days: a qualitative study. Int J Nurs Stud. 2015 Jan;52(1):288-96. doi: 10.1016/j.ijnurstu.2014.09.009. Epub 2014 Oct 5. PMID 25445033
- [Background] Lyu XC, Jiang HJ, Lee LH, Yang CI, Sun XY. Oncology nurses' experiences of providing emotional support for cancer patients: a qualitative study. BMC Nurs. 2024 Jan 20;23(1):58. doi: 10.1186/s12912-024-01718-1. PMID 38245735
- [Background] Kostka AM, Borodzicz A, Krzeminska SA. Feelings and Emotions of Nurses Related to Dying and Death of Patients - A Pilot Study. Psychol Res Behav Manag. 2021 Jun 4;14:705-717. doi: 10.2147/PRBM.S311996. eCollection 2021. PMID 34113186
- [Background] Cotter P, Holden A, Johnson C, Noakes S, Urch C, King A. Coping With the Emotional Impact of Working in Cancer Care: The Importance of Team Working and Collective Processing. Front Psychol. 2022 Jul 15;13:877938. doi: 10.3389/fpsyg.2022.877938. eCollection 2022. PMID 35911049